CLINICAL TRIAL: NCT06708455
Title: Phase 2 Trial of Autologous Rapamycin-Resistant Th1/Tc1 (RAPA-201) Cell Therapy of PD-(L)1 Resistant Malignant Melanoma
Brief Title: Phase 2b of RAPA-201 Cell Therapy in Post-PD-(L)-1 Melanoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rapa Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAPA-201-MEL-PH2-01
Record Dates: First submitted 2024-11-19; First posted 2024-11-27 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Malignant Melanoma With Metastasis; Malignant Melanoma; Malignant Melanoma Stage IIIc; Malignant Melanoma Stage IV
Keywords: Adoptive T Cell Therapy; Rapamycin; Regenerative Medicine; Malignant Malanoma; RMAT
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Administration of RAPA-201 cells (Experimental): RAPA-201 cells will be administered at a target flat dose between 80 and 400 x 10^6 cells per infusion.
  Interventions: Biological: RAPA-201 Rapamycin Resistant T Cells; Drug: Chemotherapy Prior to RAPA-201 Therapy

INTERVENTIONS:
Biological: RAPA-201 Rapamycin Resistant T Cells — Autologous Rapamycin-Resistant Th1/Tc1 Cells
Drug: Chemotherapy Prior to RAPA-201 Therapy — Carboplatin + Paclitaxel Regimen (CP Regimen)

SUMMARY:
The protocol is a Simon's 2-stage, non-randomized, open label, multi-site, phase 2 trial for patients with advanced metastatic, recurrent and unresectable malignant melanoma that has recurred or relapsed after prior anti-PD-(L)1 therapy.

DETAILED DESCRIPTION:
The therapy of solid tumors, including melanoma, has been revolutionized by immune therapy, in particular, approaches that activate immune T cells in a polyclonal manner through blockade of checkpoint pathways such as the PD-1/PD-L1 pathway [PD-(L)1] by administration of monoclonal antibodies. In this study, we will evaluate the adoptive transfer of RAPA-201 cells, which are checkpoint-deficient polyclonal T cells that represent an analogous yet distinct immune therapy treatment platform for the therapy of malignant melanoma that is refractory to anti-PD-(L)1 therapy.

RAPA-201 is a second-generation immunotherapy product consisting of epigenetically reprogrammed autologous CD4+ and CD8+ T cells of Th1/Tc1 cytokine phenotype. RAPA-201, which is safely administered exclusively in the outpatient setting, is currently being evaluated for the therapy of solid tumors that are refractory to anti-PD-(L)1 therapy (NCT05144698), with accrued patients having diagnoses of non-small cell lung cancer, small cell lung cancer, squamous cell head and neck and cancer, gastric cancer, esophageal cancer, and melanoma. Because RAPA-201 is a polyclonal T cell therapy that targets potential tumor antigens in vivo, RAPA-201 may also be applicable for the therapy of other immune sensitive tumors, including but not limited to lung cancer, bladder cancer, and renal cell carcinoma.

Initial results on the first RAPA-201 clinical trial in solid tumors (NCT05144698) demonstrated that six out of 10 evaluable melanoma patients (60%) responded to RAPA-201 therapy, thus providing a rationale for this phase 2b clinical trial that will focus exclusively upon the treatment of PD-(L)1 refractory malignant melanoma. On the basis of these results, RAPA-201 therapy of treatment-refractory metastatic melanoma was granted the Regenerative Medicine Advanced Therapy (RMAT) designation by the US FDA.

The novel RAPA-201 manufacturing platform, which incorporates both an inhibitor of the mechanistic target of rapamycin (mTOR; temsirolimus) and an anti-cancer Th1/Tc1 polarizing agent (IFN-alpha) generates polyclonal T cells with five key characteristics:

1. Th1/Tc1: polarization to anti-cancer Th1 and Tc1 subsets, with commensurate down-regulation of immune suppressive Th2 and regulatory T (TREG) subsets;
2. T Central Memory: expression of a T central memory (TCM) phenotype, which promotes T cell engraftment and persistence for prolonged anti-tumor effects;
3. Rapamycin-Resistance: which translates into a multi-faceted anti-apoptotic phenotype that improves T cell fitness in the stringent conditions of the tumor microenvironment; the resistant phenotype of RAPA-201 also permits concomitant therapy with cytotoxic chemotherapy, including the outpatient carboplatin plus paclitaxel regimen utilized on this protocol or planned combination therapy with tumor targeted antibody drug conjugates (ADCs);
4. T Cell Quiescence: reduced T cell activation, as evidence by reduced expression of the IL-2 receptor CD25, which reduces T cell-mediated cytokine toxicities such as cytokine-release syndrome (CRS) that limit other forms of T cell therapy; and
5. Reduced Checkpoints: multiple checkpoint inhibitory receptors are markedly reduced on RAPA-201 cells (including but not limited to PD-1, CTLA4, TIM-3, LAG3, and LAIR1), which increases T cell immunity in the checkpoint-replete, immune suppressive tumor microenvironment; RAPA-201 follows the normal rules of immunology, with eventual checkpoint expression after RAPA-201 maturation from a TCM phenotype towards a T effector memory phenotype; because of this biology, we envision that RAPA-201 will be favorably incorporated into anti-PD-(L)1 containing combination regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 and an estimated life expectancy of ≥ 3 months.
3. Patients with unresectable or metastatic melanoma (Stage IIIc or Stage IV).
4. Prior to enrollment, documented refractory status to the most recent regimen, which must include an anti-PD-(L)1 monoclonal antibody, as defined by lack of response after at least two cycles of therapy or relapse within 12-months of initiation of the anti-PD- (L)1-containing therapy.
5. For patients with BRAF V600 mutation-positive tumors, prior therapy with a BRAF inhibitor alone or in combination with a MEK inhibitor.
6. Presence of measurable disease to permit monitoring by iRECISTv1.1 Criteria.
7. Must have a potential source of autologous T cells potentially sufficient to manufacture RAPA-201 cells, as defined by a circulating absolute lymphocyte count (ALC) of ≥ 500 cells/μL.
8. Patients must be ≥ two weeks from last solid tumor cancer chemotherapy, major surgery, radiation therapy and/or participation in investigational trials.
9. Patients must have recovered from clinical immunotherapy-related toxicities [resolution of CTCAE (v5) toxicity to a value of ≤ 1; with the exception of alopecia, vitiligo, and endocrinopathy stable on hormone replacement].
10. Hematologic parameters of: Absolute neutrophil count (ANC) of ≥ 1500 cells/μL, Platelet count ≥ 100,000 cells/μL, and Hemoglobin of ≥ 9 grams/μL.
11. Calculated creatinine clearance of ≥ 40 mL/min.
12. Ejection fraction (EF) by MUGA or 2-D echocardiogram within institution normal limits, with an EF level of ≥ 45%.
13. Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 3 x upper limit of normal (ULN) (or ≤ ULN if patient has liver metastasis).
14. Bilirubin ≤ 2.0 mg/dL (if Gilbert's disease, ≤ 3.0 mg/dL).
15. No history of abnormal bleeding tendency (as defined by any inherited coagulation defect or history of internal bleeding).
16. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

Exclusion Criteria

1. Other active malignancy (except non-melanoma skin cancer).
2. Life expectancy < 3 months.
3. Seropositivity for HIV, hepatitis B, or hepatitis C, unless such conditions are in stable condition using adequate treatment.
4. Uncontrolled hypertension.
5. Cerebrovascular accident within 6 months of enrollment.
6. Myocardial infarction within 6 months of enrollment.
7. NYHA class III/IV congestive heart failure.
8. Uncontrolled angina/ischemic heart disease.
9. Cancer metastasis to the central nervous system, unless such metastasis has been adequately treated.
10. Pregnant or breastfeeding patients.
11. Women of childbearing potential, or males who have a partner of childbearing potential, who are unwilling to practice contraception.
12. Patients may be excluded at the discretion of the PI or if it is deemed that allowing participation would represent an unacceptable medical or psychiatric risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of RAPA-201 Cell Therapy | 18 months (6 mo. of treatment; 12 mo of clinical follow-up)
  In an intent-to-treat (ITT) manner, the efficacy of RAPA-201 cell therapy will be determined by overall response rate (ORR) in metastatic melanoma patients with progressive disease after anti-PD-(L)1 therapy, as assessed by the independent review committee (IRC) per iRECIST v1.1.

SECONDARY OUTCOMES:
Characterize RAPA-201 Efficacy | One (1) year after the last dose of RAPA-201 cells.
  To further characterize RAPA-201 efficacy by measurement of duration of response (DOR; as measured in days), disease-control-rate (DCR; as measured in days ), progression-free-survival (PFS), and overall survival (OS; as measured in days), as assessed by the IRC and Site Investigator (iRECIST v1.1).
Safety of RAPA-201 Cell Therapy | One (1) year after the last dose of RAPA-201 cells.
  Safety, as measured by determination of the number and grade of any adverse event attributable to the RAPA-201 Investigational Product [using the CTCAE v4.0 nomenclature]
Quality of Life (QOL) | One (1) year after the last dose of RAPA-201 cells.
  To evaluate effect of therapy on quality of life (QOL) using the Short Form-36 Survey. The Short-Form 36 Survey that will be utilized uses a scale of 0-to-100, with higher scores indicating a better outcome.

OTHER OUTCOMES:
Immune Reconstitution | One (1) year after the last dose of RAPA-201 cells.
  To characterize the immune reconstitution pattern in recipients of RAPA-201 therapy to better understand the therapeutic mechanism and lead to biomarker or predictive tests. Immune reconstitution will be quantified by determination of the absolute lymphocyte count (ALC) at the time of study entry, after RAPA-201 therapy, and then at the patient's last study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Fowler, M.D., Study Director — Rapa Therapeutics
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States